CLINICAL TRIAL: NCT02294812
Title: Effects of Cognitive Training on Age-Related Hearing Loss and Speech Perception
Brief Title: Effects of Cognitive Training on Speech Perception
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding and staff to conduct the study
Sponsor: Aaron Newman (Other)
Responsible Party: Sponsor-Investigator, Aaron Newman, Neuropsychologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCIL-HL-CT
Record Dates: First submitted 2014-11-03; First posted 2014-11-19 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hearing Loss; Deafness and Auditory Perception
Keywords: Hearing Loss; Speech Perception; Cognitive Training; Cognitive Fitness; Memory, Short-Term
MeSH Terms: conditions — Hearing Loss; Deafness | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control, cognitive training (Active Comparator): Participants in the control arm will receive cognitive training for cognitive abilities not affected by age-related hearing loss.
  Interventions: Behavioral: Cognitive training
- Experimental, cognitive training (Experimental): Participants in the experimental arm will receive cognitive training for cognitive abilities affected by age-related hearing loss.
  Interventions: Behavioral: Cognitive training
- Active Control, crossword training (Active Comparator): Participants in this group will undergo crossword puzzle training. The purpose of this group is control for any effects that may be due to engaging in cognitive training.
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Behavioral: Cognitive training — Participants will engage in eight weeks of training that focuses on improving various cognitive abilities. For example, short term memory.
  Cognitive training will take place 30 minutes per day, five days per week, for eight weeks. Training will be done in the participant's own home using web-based software. Participants will be randomly assigned to either the active control group, the control cognitive training group, or the experimental cognitive training group following the second study visit.
  After eight weeks, participants will no longer partake in training.

SUMMARY:
In this study, the investigators are testing whether cognitive training can lead to improvements in speech perception for individuals with hearing loss. Individuals will complete 20 hours of cognitive training that is designed to improve cognitive abilities such as short term memory and attention. The investigators predict that cognitive training that improves the cognitive abilities affected by hearing loss will improve speech perception.

ELIGIBILITY:
Inclusion Criteria:

* Able to come to Dalhousie University, Halifax, Nova Scotia, Canada for study visits
* Adults (50 years or older) with mild to moderate hearing loss
* Access to an internet-connected device that is able to use Flash media, basic computer skills
* Medically stable participants
* Not currently taking medication that may affect brain function (e.g., anti-anxiety medication)
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Participants with neurological conditions such as epilepsy or concussions will be excluded for safety reasons
* Participants who are not native English speakers (materials used in the study are only in English)
* Participants who are unable to provide consent
* Participants with impaired cognition (assessed with the Montreal Cognitive Assessment)
* Participants with high accuracy on the Speech Perception in Noise task at the second study visit (to eliminate participants who may be performing at ceiling level)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Speech Perception in Noise Test - Improvement in speech perception accuracy from baseline to post-training for high and low predictability sentences | Baseline, Weeks 2, 10, and 18
  Sentences of high predictability and low predictability are played with multi-user talker babble. Participants must repeat the last word of each sentence as they heard it. The primary outcome measure will be the accuracy for repeating the sentence.

SECONDARY OUTCOMES:
Working Memory Cognitive Training - Improvements in working memory abilities from baseline | Weeks 2, 10, and 18
  Individuals are asked to participate in 20 hours of cognitive training that will focus on either improving abilities affected by hearing loss (i.e., verbal working memory), or abilities not affected by hearing loss (i.e., spatial working memory).
  Performance on the working memory task, Operation Span Task (OSPAN), will be assessed using the total score which is calculated as a sum based on the number of correct answers (letters accurately sequentially recalled) within a block for the duration of the task. Higher scores indicate better working memory capacity. Performance on the working memory cognitive training games will be assessed using the participant's accuracy, reaction time, and final score on the game.
  Improvements in working memory will be assessed by comparing participant performance on working memory tasks (OSPAN; cognitive training memory games) before receiving cognitive training, immediately after receiving cognitive training, and eight weeks post-training.
Brain Performance Test | Weeks 2 and 10
  The Brain Performance Test (BPT) is an assessment tool available online through the training program website. Participants will be assessed at home on their initial performance for a variety of cognitive abilities including stop-signal tasks, grammatical reasoning, and memory spans. After completing the eight weeks of cognitive training, participants will again be assessed at home with the BPT to determine whether there are any improvements in cognitive abilities.
Attention Cognitive Training - Improvements in attention abilities from baseline | Weeks 2, 10, and 18
  Individuals are asked to participate in 20 hours of cognitive training. Cognitive training will focus on either improving abilities affected by hearing loss (i.e., attention), or abilities not affected by hearing loss (i.e., spatial working memory).
  Performance on the attention task, Flanker-Simon, will be assessed based on participant's accuracy and reaction time for the Flanker task, and the Simon task.
  Performance on the attention cognitive training games will be assessed using the participant's accuracy, reaction time, and final score on the game.
  Improvements in attention will be assessed by comparing the performance of participants on attention tasks (Flanker-Simon; cognitive training attention games) before receiving cognitive training, immediately after receiving cognitive training, and eight weeks post-training.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Newman, PhD, Principal Investigator — Dalhousie University, Canada
Locations (1):
- NeuroCognitive Imaging Lab, Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NeuroCognitive Imaging Lab — http://www.ncilab.ca/